CLINICAL TRIAL: NCT03795558
Title: A Study to Investigate the Influence of PTH-lowering by Etelcalcetide (Parsabiv®) on the Calcification Propensity of Serum in Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prim. Priv. Doz. Dr. Daniel Cejka (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Prim. Priv. Doz. Dr. Daniel Cejka, Head of Nephrology department, Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Etelcalcetide-T50-CKD5D
Record Dates: First submitted 2018-09-18; First posted 2019-01-07 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, dose-escalation, pilot study. Starting dose 2.5 mg thrice weekly dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Etelcalcetide 2.5 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide
- Etelcalcetide 5 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide
- Etelcalcetide 7,5 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide
- Etelcalcetide 10 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide
- Etelcalcetide 12,5 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide
- Etelcalcetide 15 mg (Experimental): Etelcalcetide, starting dose of 2.5mg thrice weekly, dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Up-Titration
  Other Names: Parsabiv

SUMMARY:
This is a single-center, prospective, dose-escalation, pilot study in 15 end-stage renal disease patients on chronic hemodialysis with secondary hyperparathyroidism.

DETAILED DESCRIPTION:
Fifteen prevalent and stable hemodialysis patients with secondary hyperparathyroidism eligible for treatment with calcium receptor sensitizers according to current KDIGO will be included.

Study phases will begin and end on the day of the first hemodialysis session of the week.

The run-in phase will last 4 weeks. No calcimimetics will be prescribed during the run-in phase.

The treatment phase starts with a dose of etelcalcetide is 2.5mg thrice weekly. Etelcalcetide dose will be escalated every 4 weeks in 2.5mg/dialysis session increments to a maximum dose of 15mg thrice weekly.

The wash-out Phase starts after completion of the 15mg thrice-weekly phase or in case a pre-specified safety endpoint is reached, etelcalcetide will be discontinued and patients will be followed for additional 8 weeks to study any potential reversibility of PTH lowering on T50 results.

For the individual patient, the study duration will be 9 months

ELIGIBILITY:
Inclusion Criteria:

* Prevalent patients (≥ 3 months on dialysis) treated with thrice weekly hemodialysis (HD) or hemodiafiltration (HDF)
* Secondary hyperparathyroidism defined as PTH levels > 9x ULN according to current KDIGO guidelines if therapy-naïve, or patients already treated with calcium receptor sensitizers with PTH > 2x ULN
* Albumin corrected calcium ≥ 2,08 mmol/l
* Calcium concentrations of dialysate stable for at least 2 weeks prior to screening

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study or participation in non-interventional studies
* Current treatment with etelcalcetide (Parsabiv©) or treatment with etelcalcetide within 3 months prior to study inclusion
* Patient has known sensitivity to any of the products or components of Parsabiv©
* Patient has received a parathyroidectomy
* Parathyroidectomy planned or expected during the study period
* Elective kidney transplant scheduled during the study period
* Therapy with bisphosphonates within the past 12 months
* Therapy with denosumab within the past 6 months
* Antacids containing aluminum, calcium, magnesium or bicarbonate
* Patient has a history of symptomatic ventricular arrhythmias or Torsades de Pointes
* Patient has a history of myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 6 months prior to screening.
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
T50-Laboratory Test for measuring calcification | 32 weeks
  The changes in T50 values between the different study phases will be evaluated as the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cejka, Md, Principal Investigator — Head of Nephrology
Locations (1):
- Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria, Austria